CLINICAL TRIAL: NCT07024680
Title: Real World Study of Effectiveness of Sunitinib or Sorafenib as First Line Therapy to Chinese Unresectable Locally Advanced or Metastatic Papillary Renal Cell Carcinoma: a Multi-center, Retrospective, Observational Study
Brief Title: Real World Study of Effectiveness of Sunitinib or Sorafenib to Chinese Unresectable Locally Advanced or Metastatic PRCC
Acronym: PRCC
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5086R00001
Record Dates: First submitted 2025-03-21; First posted 2025-06-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Papillary Renal Cell Carcinoma
Keywords: papillary renal cell carcinoma;; sunitinib;; sorafenib;; real world study.
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- unresectable locally advanced or metastatic papillary renal cell carcinoma: unresectable locally advanced or metastatic papillary renal cell carcinoma
  Interventions: Other: Observational, None intervention

INTERVENTIONS:
Other: Observational, None intervention — Observational, None intervention

SUMMARY:
This is a multi-center, observational, retrospective study designed to characterize the effectiveness and safety of sunitinib or sorafenib monotherapy in the treatment of Chinese adult patients with unresectable and locally advanced or metastatic PRCC, who have not received any prior systemic anticancer therapy in the metastatic setting. Electronic medical record (EMR) data of patients with 1L sunitinib or sorafenib monotherapy will be screened from Grade-A Tertiary hospitals in China. The study period is from 1st September 2007 to 31st December 2024.

DETAILED DESCRIPTION:
This is a multi-center, observational, retrospective study designed to characterize the effectiveness and safety of sunitinib or sorafenib monotherapy in the treatment of Chinese adult patients with unresectable and locally advanced or metastatic PRCC, who have not received any prior systemic anticancer therapy in the metastatic setting.

Data will be screened and collected from Grade-A Tertiary hospitals in different provinces across China. Relevant patient-level information will be screened from EMR in multiple information systems in these hospitals. Information on baseline covariates, exposures and outcomes will be collected from hospital, including laboratory results, radiology and pathology reports, physician and nurse notes, prescriptions written and dispensed, surgical procedures, primary and subsequent diagnoses, and other details of a patient's outpatient visits and hospital admissions. Patients' information data will be collected and entered into the electronic data capture (EDC) system.

The study population consist of unresectable and locally advanced or metastatic PRCC patients in China who received 1L sunitinib or sorafenib between 1st September 2007 and 30th June 2024. Patients who were initially diagnosed with early stage PRCC and whose disease later progressed to unresectable and locally advanced or metastatic PRCC are eligible to be included in the study. Moreover, patients who relapsed after nephrectomy are also eligible to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be included in the real-world cohort:

1. Age ≥ 18 years at the index date
2. One of the following:

1)diagnosed with unresectable and locally advanced, or metastatic PRCC; 2)diagnosed with unresectable and locally advanced, or metastatic RCC, and with papillary (papillary ≥ 50%) as the dominant and presumed primary histology type.

3.Patients who received 1L therapy of sunitinib or sorafenib 4.Patients with tumor assessment or relevant clinical visit within 6-month follow-up since index date. (The rationale and details of 6-month minimal follow-up is presented in section 3.6). Death events within 6-month will be included.

Exclusion Criteria:

Patients who meet one or more following criteria will be excluded from the real-world cohort:

1. Patients with papillary urothelial carcinoma or renal pelvis cancer of the kidney;
2. Patients with history of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 5 years;
3. Patients who received systemic anti-cancer therapy for PRCC prior to the index date; The following is exception:

   Prior systemic anti-cancer therapy in the neoadjuvant or adjuvant setting are acceptable if it was completed more than 12 months before metastatic/recurrent disease was diagnosed.

   For patients who received prior systemic neoadjuvant/adjuvant therapies within 12 months before metastatic/recurrent disease was diagnosed, the neoadjuvant/adjuvant therapy will be counted as 1L therapy.

   Patients are deemed eligible if the first therapy was only sustained for ≤ 3 days.
4. Patients with missing both day and month of index date;
5. Patients with severe conditions that are greater or equal to grade 3 by the definition of CTCAE 5.0 criteria when included into the study;
6. Patients who treated with any combination of chemotherapy, targeted therapy, or immunotherapy with sunitinib or sorafenib as 1L therapy.

Other exclusion criteria revised according to study D5086C00001 (SAMETA) will also be applied, only if explicit evidence can be identified in the EMR data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unresectable locally advanced or metastatic papillary renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-07-14 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to characterize the real-world PFS (rwPFS) with either sunitinib or sorafenib. | at least 6 months
  The rwPFS is defined as time from the initiation of first dose of sunitinib or sorafenib until investigator-reported disease progression (assessed by physician's notes or radiology report), or death due to any cause (in the absence of progression), whichever occurred first.

SECONDARY OUTCOMES:
The secondary objective is to characterize the rwPFS with sunitinib. | at least 6 months
  The rwPFS is defined as time from the initiation of first dose of sunitinib until investigator-reported disease progression (assessed by physician's notes or radiology report), or death due to any cause (in the absence of progression), whichever occurred first.

OTHER OUTCOMES:
To characterize the OS with either sunitinib or sorafenib monotherapy | at least 6 months
  OS is defined as time from initiation of sunitinib or sorafenib until the date of death due to any cause.
To characterize the real-world ORR (rwORR) with either sunitinib or sorafenib monotherapy | at least 6 months
  The measure of interest is rwORR, defined as the proportion of participants who have reached CR or PR as determined by investigator-reported assessment.
To characterize the time-to-treatment discontinuation (TTD) with either sunitinib or sorafenib monotherapy | at least 6 months
  The TTD is defined as time from the date of initiation of sunitinib or sorafenib till their discontinuation due to any reasons or death.
To characterize the OS with sunitinib monotherapy. | at least 6 months
  OS is defined as time from initiation of sunitinib until the date of death due to any cause.
To characterize the rwORR with sunitinib monotherapy. | at least 6 months
  The measure of interest is rwORR, defined as the proportion of participants who have reached CR or PR as determined by investigator-reported assessment.
To characterize the TTD with sunitinib monotherapy. | at least 6 months
  The TTD is defined as time from the date of initiation of sunitinib till its discontinuation due to any reasons or death.
To characterize the rwPFS with sorafenib monotherapy. | at least 6 months
  The rwPFS is defined as time from the initiation of first dose of sorafenib until investigator-reported disease progression, or death due to any cause, whichever occurred first.
To characterize the OS with sorafenib monotherapy. | at least 6 months
  OS is defined as time from initiation of sorafenib until the date of death due to any cause.
To characterize the rwORR with sorafenib monotherapy. | at least 6 months
  The measure of interest is rwORR, defined as the proportion of participants who have reached CR or PR as determined by investigator-reported assessment.
To characterize the TTD with sorafenib monotherapy. | at least 6 months
  The TTD is defined as time from the date of initiation of sorafenib till its discontinuation due to any reasons or death.
To describe the adverse events (AEs) in Chinese patients of locally advanced or metastatic PRCC treated with either sunitinib or sorafenib monotherapy/ treated with sunitinib monotherapy/ treated with sorafenib monotherapy | at least 6 months
  AEs will be evaluated in terms of:
  Occurrence and frequency Seriousness AE with outcome of death AEs leading to discontinuation of sunitinib or sorafenib

CONTACTS AND LOCATIONS:
Overall Officials: DingWei Ye, Postdoctoral, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No